CLINICAL TRIAL: NCT02679443
Title: Optimum Duration of Vitamin B12 and Folate Supplementation in Non-squamous Non-small Cell Lung Cancer (NSCLC) Patients Undergoing Pemetrexed Containing Chemotherapy: a Randomized Controlled Trial
Brief Title: Vitamin Supplementation in NSCLC Patients on Pemetrexed Based Chemotherapy
Acronym: PEMVITASTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Navneet Singh, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NK/2376/DM/913
Record Dates: First submitted 2016-02-01; First posted 2016-02-10 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Lung Adenocarcinoma; Neutropenia; Anemia; Thrombocytopenia; Nonsquamous Nonsmall Cell Neoplasm of Lung
Keywords: Lung Adenocarcinoma; Non-squamous NSCLC; Chemotherapy; Pemetrexed; Vitamin B12; Folate; Supplementation; Cytopenia
MeSH Terms: conditions — Adenocarcinoma of Lung; Neutropenia; Anemia; Thrombocytopenia; Cytopenia | interventions — Folic Acid; Vitamin B 12

ARMS (2):
- Delayed Arm (No Intervention): Participants are started on folate and vitamin B12 supplementation for 5-7 days prior to initiation of chemotherapy
- Immediate Arm (Experimental): Participants are started on folate and vitamin B12 supplementation simultaneously with chemotherapy (within 24 hours of initiation of chemotherapy)
  Interventions: Dietary Supplement: Folate and B12

INTERVENTIONS:
Dietary Supplement: Folate and B12 — Vitamin (folate and B12) supplementation started simultaneously with initiation of chemotherapy (within 24 hours of initiation of chemotherapy). The only difference from the delayed (no-intervention) arm is the timing of initiation of vitamin supplementation. Dose and mode of administration of vitamin B12 and folate supplementation remain similar in both arms.
  Arms: Immediate Arm

SUMMARY:
Folic acid (FA; folate) in the dose of 350-1,000 μg daily should be supplemented, daily, starting 7 days before the first dose of pemetrexed based chemotherapy and should be continued while the patient is on therapy and for 21 days after cessation of therapy. Vitamin B12 injections (1,000 μg i.m.) should also be started 1 week before the first dose of chemotherapy. However, the evidence for delaying chemotherapy by seven days for the purpose of giving vitamin B12 and FA supplementation is not robust. Observational and prospective single arm studies have not shown any increased toxicity if pemetrexed was started earlier than the recommended duration of supplementation. In a resource constrained setting, this will lead to one additional visit and 1-week chemotherapy delay which may be inconvenient for patients.

Hence an open label, randomized control trial is being undertaken to evaluate if there are any differences in pemetrexed related hematological toxicity amongst patients who receive delayed initiation of chemotherapy (following 5 - 7 days of vitamin B12 and FA supplementation; Delayed Arm) as compared to those in whom vitamin B12 and FA supplementation is starting simultaneously (within 24 hours) of initiation of chemotherapy (Immediate Arm).

DETAILED DESCRIPTION:
Chemotherapy Regimen:

All patients will receive pemetrexed and cisplatin in doses of 500 mg and 65 mg, respectively, per square meter of body surface area each on day 1 of a 3-week cycle. Patients with contraindications to administration of cisplatin, those who are intolerant to cisplatin, or develop grade 3 or 4 adverse events from cisplatin will be given carboplatin in combination with pemetrexed. Carboplatin will be given at a dose calculated to produce an area under the concentration-time curve (AUC) of 5.0mg/mL/min. Dose modifications of either pemetrexed or the platinum agent or both will be done in case of significant change in PS or toxicity from or intolerance to dose administered in the previous cycle.

Supplementation:

1. Folic acid (FA) supplementation will be given to all patients orally in the dose of 5 ml (1000 μg) once daily of VITCOFOL (FDC Limited, Mumbai, India) pediatric formulation, which contains 200 μg FA/ml of the preparation. Patients will be instructed to measure the prescribed dose using a 5 ml plastic syringe containing markings at every 0.5 ml. Patients will also be instructed not to take any additional multivitamin supplements. In addition to FA supplementation, all patients will also be started simultaneously on oral iron (ferrous sulphate 200 mg twice a day). Once initiated, both FA and ferrous sulphate will be given on a daily basis and continued throughout the duration of chemotherapy and for at least 3 weeks beyond the last cycle.
2. Vitamin B12 supplementation will be given to all patients intramuscularly in the dose of 1000 μg along with each cycle of chemotherapy (maximum of six doses during the study period).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic (Stage IIIB/IV) NSCLC and Stage III A NSCLC, not scheduled for upfront surgical resection
* Nonsquamous histology (including adenocarcinoma)
* At least one unidimensionally measurable lesion, according to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.0), or at least one nonmeasurable lesion that was assessable using conventional techniques or a spiral computed tomography scan
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* No previous chemotherapy for advanced disease and no previous targeted molecular therapy
* Adequate liver and renal function;
* Previous radiation therapy is permitted if completed >4 weeks before enrollment and the patient has recovered from any treatment-related toxicity.

Exclusion Criteria:

* Hemoglobin value < 9gm/dl
* Required erythropoiesis stimulating agents or blood transfusions in the recent past (4 months)
* Symptomatic untreated brain metastasis
* Any previous malignancy
* Concurrent use of any other tumor therapy
* Active infection or a serious concomitant disorder
* Inability to interrupt nonsteroidal anti-inflammatory agents
* Inability or unwillingness to take folic acid, vitamin B12, or dexamethasone supplementation
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of any grade hematological toxicity | Completion of six cycles (average of 18 weeks; each cycle is 21 days) of pemetrexed-platinum doublet chemotherapy
  Incidence of Grade 1-5 Anemia, Grade 1-5 Neutropenia, Grade 1-5 Thrombocytopenia (all graded according to NCI CTCAE Version 3.0) related to pemetrexed-platinum doublet chemotherapy during the study period

SECONDARY OUTCOMES:
Incidence of grade 3/4 hematological toxicity | Completion of six cycles (average of 18 weeks; each cycle is 21 days) of pemetrexed-platinum doublet chemotherapy
  Incidence of Grade 3-4 Anemia, Grade 3-4 Neutropenia, Grade 3-4 Thrombocytopenia (all graded according to NCI CTCAE Version 3.0) related to pemetrexed-platinum doublet chemotherapy during the study period
Number of doses of G-CSF administered | Completion of six cycles (average of 18 weeks; each cycle is 21 days) of pemetrexed-platinum doublet chemotherapy
  Number of doses of G-CSF (granulocyte colony stimulating factor) administered during the study period
Number of doses of ESAs administered | Completion of six cycles (average of 18 weeks; each cycle is 21 days) of pemetrexed-platinum doublet chemotherapy
  Number of doses of ESAs (erythropoiesis stimulating agents) administered during the study period
Number of PRBC transfusions administered | Completion of six cycles (average of 18 weeks; each cycle is 21 days) of pemetrexed-platinum doublet chemotherapy
  Number of PRBC (packed red blood cell) transfusions administered during the study period
Relative Dose Intensity (RDI) delivered | Completion of six cycles (average of 18 weeks; each cycle is 21 days) of pemetrexed-platinum doublet chemotherapy
  RDI (in percentage) will be calculated as [(delivered dosage/predicted dosage)*100]. This will be calculated separately for pemetrexed and platinum compounds for each chemotherapy cycle and also averaged for the total duration of chemotherapy
Number of Inter-Cycle Delays (ICDs) | Completion of six cycles (average of 18 weeks; each cycle is 21 days) of pemetrexed-platinum doublet chemotherapy
  ICD will be defined as a delay of at least 7 days between scheduled date and actual date of administration of a given cycle of chemotherapy

OTHER OUTCOMES:
Changes in serum levels of folic acid and homocysteine | Completion of six cycles (average of 18 weeks; each cycle is 21 days) of pemetrexed-platinum doublet chemotherapy
  After third and after sixth cycle of pemetrexed-platinum doublet chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Navneet Singh, MD DM, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

REFERENCES:
- [Derived] Singh N, Baldi M, Kaur J, Muthu V, Prasad KT, Behera D, Bal A, Gupta N, Kapoor R. Timing of folic acid/vitamin B12 supplementation and hematologic toxicity during first-line treatment of patients with nonsquamous non-small cell lung cancer using pemetrexed-based chemotherapy: The PEMVITASTART randomized trial. Cancer. 2019 Jul 1;125(13):2203-2212. doi: 10.1002/cncr.32028. Epub 2019 Mar 2. PMID 30825389
- [Derived] Baldi M, Behera D, Kaur J, Kapoor R, Singh N. Rationale and Design of PEMVITASTART-An Open-label Randomized Trial Comparing Simultaneous Versus Standard Initiation of Vitamin B12 and Folate Supplementation in Nonsquamous, Non-Small-cell Lung Cancer Patients Undergoing First-line Pemetrexed-based Chemotherapy. Clin Lung Cancer. 2017 Jul;18(4):432-435. doi: 10.1016/j.cllc.2016.11.017. Epub 2016 Dec 2. PMID 28073680